CLINICAL TRIAL: NCT01720914
Title: Instruments for Delirium Assessment Regarding to Analgesia Sedation and Ventilator Status
Acronym: IDEAS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: IDEAS
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patient

SUMMARY:
In this prospective, multicenter observational study we assess the diagnostic validity of the following standard screening instruments for delirium regarding sedation, analgesia and ventilator status in critically ill patients:

* Confusion Assessment Method for the ICU (CAM-ICU)
* Intensive Care Delirium Screening Checklist (ICDSC)
* Nursing-Delirium-Screening-Scale (Nu-DESC)

The definite delirium diagnosis (definite in terms of reference standard) is made according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders 4th Edition, text revised (DSM-IV-TR) published by the American Psychiatric Association (APA) which is the Gold Standard to diagnose delirium.

Primary research question: Does sedation, ventilator status and analgesia influence the sensitivity of delirium screening tools (DST)?

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patient
* Patient age > 18 years

Exclusion Criteria:

* Neurosurgical patients
* Severe brain injury, intracerebral bleeding, stroke
* Inability to communicate due to anacusia or severe hearing loss
* Insufficient language comprehension
* Patients < 24 h total time of Intensive Care Unit stay
* Deep sedation (RASS < -3) for ≥ 7 days during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult critically ill patients
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the delirium screening/diagnosing tool "Confusion Assessment Method for the ICU (CAM-ICU)" regarding sedation and ventilator status. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV TR criteria
Sensitivity of the delirium-screening tool "Intensive-Care Delirium Screening Checklist(ICDSC)" regarding sedation and ventilator status. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV TR criteria.
Sensitivity of the delirium screening tool "Nursing Delirium Screening Scale (Nu-DESC)" regarding sedation and ventilator status. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV TR criteria

SECONDARY OUTCOMES:
Specificity of the "Confusion Assessment Method for the ICU (CAM-ICU)", the "Intensive Care Delirium Screening Checklist (ICDSC)" and the "Nursing Delirium Screening Scale" regarding sedation and ventilator status. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV-TR criteria.
Calculation and Analysis of the positive predictive values of the assessed delirium-screening scales. | Participants will be followed in the 7-days sample period
  Calculation of positive and negative predictive values of the "Confusion Assessment Method for the ICU (CAM-ICU)", the "Intensive Care Delirium Screening Checklist (ICDSC)" and the "Nursing Delirium Screening Scale" regarding sedation and ventilator status.
  Used reference standard: DSM-IV-TR criteria
Incidence of delirium | Participants will be followed in the 7-days sample period
  According to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and Confusion Assessment Method for the ICU (CAM-ICU)
Incidence of Subsyndromale Delirium (SSD) | Participants will be followed in the 7-days sample period
  According to Intensive Care Delirium Screening Checklist (ICDSC) and Nursing Delirium Screening Scale (Nu-DESC)
Analgesia | Participants will be followed in the 7-days sample period:
  According to Numeric rating scale visually enlarged and laminated (NRS-V), Behavioural pain scale (BPS) and Behavioural pain scale not intubated (BPS-NI)
Ventilator status | Participants will be followed in the 7-days sample period
  Clinical observation of A) whether an airway is used B)whether a patient is ventilated with a positive pressure ventilation or a high flow ventilation for more than 6 hours per day.
Administered neuroleptics, cumulative | Participants will be followed in the 7-days sample period
Administered analgesics, cumulative | Participants will be followed in the 7-days sample period
Administered sedatives, cumulative | Participants will be followed in the 7-days sample period
Severity of illness | Participants will be followed in the 7-days sample period
  according to Acute Physiology And Chronic Health score (APACHE 2), Simplified Acute Physiology Score (SAPS 2) and Sequential Organ Failure Assessment score (SOFA)
Antibiotics/infections | Participants will be followed in the 7-days sample period
ICU length of stay | Participants will be followed for the duration of intensive care unit stay and hospital stay, an expected average of 4 weeks
Duration of mechanical ventilation | Participants will be followed for the duration of intensive care unit stay and hospital stay, an expected average of 4 weeks
Discharge mode | Participants will be followed for the duration of intensive care unit stay and hospital stay, an expected average of 4 weeks
28-day mortality | Participants will be followed for the duration of intensive care unit stay and hospital stay, an expected average of 4 weeks
Specificity of the "Confusion Assessment Method for the ICU (CAM-ICU)", the "Intensive Care Delirium Screening Checklist (ICDSC)" and the "Nursing Delirium Screening Scale" regarding analgesia. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV-TR criteria.
Sensitivity of the "Confusion Assessment Method for the ICU (CAM-ICU)", the "Intensive Care Delirium Screening Checklist (ICDSC)" and the "Nursing Delirium Screening Scale" regarding analgesia. | Participants will be followed in the 7-days sample period
  Used reference standard: DSM-IV-TR criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Centro de Terapia Intensiva da Hospital Pro-Cardiaco, Botafogo, Rio de Janeiro, Brazil
- Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité -University Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Nacul FE, Paul N, Spies CD, Sechting H, Hecht T, Dullinger JS, Piper SK, Luetz A, Balzer FS, Wernecke KD, Sa AK, Barros Ferreira da Costa C, Eymold L, Chenitir C, Weiss B. Influence of Sedation Level and Ventilation Status on the Diagnostic Validity of Delirium Screening Tools in the ICU-An International, Prospective, Bi-Center Observational Study (IDeAS). Medicina (Kaunas). 2020 Aug 13;56(8):411. doi: 10.3390/medicina56080411. PMID 32823781